CLINICAL TRIAL: NCT04040647
Title: Tolerance of Early Mobilization and Ambulation the Day of Colorectal and Bariatric Surgery in an Enhanced Recovery Program
Brief Title: Tolerance of Early Postoperative Mobilization and Ambulation
Acronym: MOBTOL
Status: Completed | Type: Observational
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Jean François Brichant, Professor in Anesthesiology, chief of service, University of Liege
Other Study IDs: 2019/MOBTOL
Record Dates: First submitted 2019-07-24; First posted 2019-08-01 (Actual); Last update posted 2020-05-14 (Actual); Status verified 2020-05

CONDITIONS: Ambulation Difficulty; Colorectal Surgery; Bariatric Surgery
MeSH Terms: conditions — Mobility Limitation | interventions — Walking

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- colorectal surgery: 50 consecutive patients scheduled to colorectal surgery in an enhanced recovery programme
  Interventions: Behavioral: mobilization and ambulation
- bariatric surgery: 50 consecutive patients scheduled to bariatric surgery (gastric by-pass, sleeve gastrectomy) in an enhanced recovery programme
  Interventions: Behavioral: mobilization and ambulation

INTERVENTIONS:
Behavioral: mobilization and ambulation — 6-min walk test (6-MWT)

SUMMARY:
Enhanced recovery programme (ERP) includes early postoperative mobilization and ambulation the day of surgery. Data suggest that orthostatic symptoms prevent a large number of patients from ambulating the day of surgery. The investigators plan to include 50 patients scheduled for colorectal surgery and bariatric surgery in an ERP. A 6-min walk test (6MWT) will be performed before surgery, 3 hour after the end of surgery, and 24 hour after surgery. The day of surgery a 2-min walk test will be realized.

DETAILED DESCRIPTION:
Enhanced recovery programme (ERP) includes early postoperative mobilization and ambulation the day of surgery. Data suggest that orthostatic symptoms prevent a large number of patients (up to 50%) from ambulating the day of surgery.

The investigators plan to include 50 patients scheduled for colorectal surgery and bariatric surgery in an ERP.

The primary endpoint will be the ability to get out of the bed and sit in an armchair. Orthostatic symptom will be recorded. The secondary endpoint will be a 6-min walk test (6-MWT). This test will be performed before surgery, 3 hour after the end of surgery, and 24 hour after surgery. The day of surgery a 2-min walk test (2-MWT) will be realized.

Correlation of the ability to early ambulate and postoperative course (adherence to ERP, complications) will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

Patients scheduled for colorectal or bariatric surgery within an ERP

Exclusion Criteria:

Patient refusal to participate, inability to walk or stand up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for colorectal or bariatric surgery within an ERP
Sampling Method: Non-Probability Sample
Enrollment: 88 (Actual)
Dates: Start 2019-09-15 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-04-01 (Actual)

PRIMARY OUTCOMES:
Number of patients with orthostatic intolerance | 24 hour after surgery
  orthostatic intolerance is defined as the occurrence of one of the following symptom when the patient stands up : presyncope, dizziness, nausea-vomiting, feeling of heat and blurred vision

SECONDARY OUTCOMES:
6-min walk test | 24 hour after surgery
  This test measures the distance covered during 6-min at normal speed

CONTACTS AND LOCATIONS:
Overall Officials: Jean L Joris, MD, Principal Investigator — Centre Hospitalier Universitaire de Liege
Locations (2):
- Belgium (2):
  - CHU Liege,, Liège
  - CHU Liege, Liège

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Eriksen JR, Munk-Madsen P, Kehlet H, Gogenur I. Orthostatic intolerance in enhanced recovery laparoscopic colorectal resection. Acta Anaesthesiol Scand. 2019 Feb;63(2):171-177. doi: 10.1111/aas.13238. Epub 2018 Aug 10. PMID 30094811
- [Result] Hanada M, Tawara Y, Miyazaki T, Sato S, Morimoto Y, Oikawa M, Niwa H, Eishi K, Nagayasu T, Eguchi S, Kozu R. Incidence of orthostatic hypotension and cardiovascular response to postoperative early mobilization in patients undergoing cardiothoracic and abdominal surgery. BMC Surg. 2017 Nov 28;17(1):111. doi: 10.1186/s12893-017-0314-y. PMID 29183368
- [Result] Skarin MU, Rice DA, McNair PJ, Kluger MT. Orthostatic intolerance following hip arthroplasty: incidence, risk factors and effect on length of stay: A prospective cohort study. Eur J Anaesthesiol. 2019 Feb;36(2):123-129. doi: 10.1097/EJA.0000000000000940. PMID 30540643